CLINICAL TRIAL: NCT04426253
Title: Identification of Genetic Factors Determining Disease Course and Preparation of Pharmacogenetic Applications in the New Type of Coronavirus Infection, COVID-19
Brief Title: Identification of Genetic Factors Determining Disease Course in the New Type of Coronavirus Infection, COVID-19
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Szeged University (Other)
Responsible Party: Sponsor
Other Study IDs: COVID19_HUNGEN_001
Record Dates: First submitted 2020-06-09; First posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: COVID-19; Sars-CoV2
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, nose and throat swab
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study aims to identify environmental factors and genetic (gene mutation and gene expression) changes, which influencing the course of the disease the new type of coronavirus infection COVID-19 in patients nationwide in a multicenter study.

At first in the study will be performed 200 patients, selected for a homogeneous groups on the basis of the patient's anamnestic data, genetic testing.

Following the interim analysis, based on the results, another 800 people are planned to involve.

ELIGIBILITY:
Inclusion Criteria:

* confirmed covid 19 infection

Exclusion Criteria:

* informed refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-06-05 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
Identification of genetic factors determining the course of the disease in case of COVID-19 | 2020. December
  Exploring genotype-phenotype connections based on anamnestic data of patients and joint bioinformatics analysis of its genetic variants

CONTACTS AND LOCATIONS:
Overall Officials: Márta Széll, MD, Ph.D., Principal Investigator — University of Szeged, Department of Medical Genetics
Locations (14):
- Hungary (14):
  - University of Pécs 1st Department of Internal Medicine Intensive Care Unit, Pécs
  - University of Pécs First Department of Internal Medicine, Pécs
  - University of Pécs Infection Department of the Coronavirus Center, Pécs
  - University of Pécs Institute of Laboratory Medicine, Pécs
  - University of Pécs Szentágotahi Research Centre, Pécs
  - University of Pécs Szentágothai Research Centre Genomics and Bioinformatics Core Facility, Pécs
  - University of Szeged Szentágothai Research Centre Virology Research Group, Pécs
  - University of Szeged Department of Anaesthesiology And Inthensive Therapy, Szeged
  - University of Szeged Department of Dermatology and Allergology, Szeged
  - University of Szeged Department of Medical Biology, Szeged
  - University of Szeged Department of Paediatrics, Szeged
  - University of Szeged First Department of Medicine, Szeged
  - University of Szeged Institute of Clinical Microbiology, Szeged
  - University of Szeged Institute of Medical Microbiology and Immunobiology, Szeged

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Danis J, Janovak L, Guban B, Goblos A, Szabo K, Kemeny L, Bata-Csorgo Z, Szell M. Differential Inflammatory-Response Kinetics of Human Keratinocytes upon Cytosolic RNA- and DNA-Fragment Induction. Int J Mol Sci. 2018 Mar 8;19(3):774. doi: 10.3390/ijms19030774. PMID 29518010
- [Background] Chiu RW, Tang NL, Hui DS, Chung GT, Chim SS, Chan KC, Sung YM, Chan LY, Tong YK, Lee WS, Chan PK, Lo YM. ACE2 gene polymorphisms do not affect outcome of severe acute respiratory syndrome. Clin Chem. 2004 Sep;50(9):1683-6. doi: 10.1373/clinchem.2004.035436. No abstract available. PMID 15331509
- [Background] Pinheiro DS, Santos RS, Jardim PCBV, Silva EG, Reis AAS, Pedrino GR, Ulhoa CJ. The combination of ACE I/D and ACE2 G8790A polymorphisms revels susceptibility to hypertension: A genetic association study in Brazilian patients. PLoS One. 2019 Aug 20;14(8):e0221248. doi: 10.1371/journal.pone.0221248. eCollection 2019. PMID 31430320
- [Background] Scepanovic P, Alanio C, Hammer C, Hodel F, Bergstedt J, Patin E, Thorball CW, Chaturvedi N, Charbit B, Abel L, Quintana-Murci L, Duffy D, Albert ML, Fellay J; Milieu Interieur Consortium. Human genetic variants and age are the strongest predictors of humoral immune responses to common pathogens and vaccines. Genome Med. 2018 Jul 27;10(1):59. doi: 10.1186/s13073-018-0568-8. PMID 30053915
- [Background] Dean L. Abacavir Therapy and HLA-B*57:01 Genotype. 2015 Sep 1 [updated 2025 Apr 21]. In: Pratt VM, Scott SA, Pirmohamed M, Esquivel B, Kattman BL, Malheiro AJ, editors. Medical Genetics Summaries [Internet]. Bethesda (MD): National Center for Biotechnology Information (US); 2012-. Available from http://www.ncbi.nlm.nih.gov/books/NBK315783/ PMID 28520363
- [Background] Danis J, Goblos A, Gal B, Sulak A, Farkas K, Torok D, Varga E, Korom I, Kemeny L, Szell M, Bata-Csorgo Z, Nagy N. Nuclear Factor kappaB Activation in a Type V Pityriasis Rubra Pilaris Patient Harboring Multiple CARD14 Variants. Front Immunol. 2018 Jul 3;9:1564. doi: 10.3389/fimmu.2018.01564. eCollection 2018. PMID 30018619
- [Background] Cao Y, Li L, Feng Z, Wan S, Huang P, Sun X, Wen F, Huang X, Ning G, Wang W. Comparative genetic analysis of the novel coronavirus (2019-nCoV/SARS-CoV-2) receptor ACE2 in different populations. Cell Discov. 2020 Feb 24;6:11. doi: 10.1038/s41421-020-0147-1. eCollection 2020. No abstract available. PMID 32133153
- [Background] Teng DH, Chen Y, Lian L, Ha PC, Tavtigian SV, Wong AK. Mutation analyses of 268 candidate genes in human tumor cell lines. Genomics. 2001 Jun 15;74(3):352-64. doi: 10.1006/geno.2001.6551. PMID 11414763
- [Background] Paoloni-Giacobino A, Chen H, Peitsch MC, Rossier C, Antonarakis SE. Cloning of the TMPRSS2 gene, which encodes a novel serine protease with transmembrane, LDLRA, and SRCR domains and maps to 21q22.3. Genomics. 1997 Sep 15;44(3):309-20. doi: 10.1006/geno.1997.4845. PMID 9325052
- [Background] Lin M, Tseng HK, Trejaut JA, Lee HL, Loo JH, Chu CC, Chen PJ, Su YW, Lim KH, Tsai ZU, Lin RY, Lin RS, Huang CH. Association of HLA class I with severe acute respiratory syndrome coronavirus infection. BMC Med Genet. 2003 Sep 12;4:9. doi: 10.1186/1471-2350-4-9. PMID 12969506
- [Background] Manczinger M, Boross G, Kemeny L, Muller V, Lenz TL, Papp B, Pal C. Pathogen diversity drives the evolution of generalist MHC-II alleles in human populations. PLoS Biol. 2019 Jan 31;17(1):e3000131. doi: 10.1371/journal.pbio.3000131. eCollection 2019 Jan. PMID 30703088
- See also: COVID-19 situation update worldwide — https://www.ecdc.europa.eu/en/geographical-distribution-2019-ncov-cases
- See also: Total Coronavirus Cases in Italy — https://www.worldometers.info/coronavirus/country/italy/
- See also: Coronavirus kills 4 family members and sickens others after a dinner in New Jersey — https://edition.cnn.com/2020/03/19/health/new-jersey-coronavirus-family-members-killed/index.html
- See also: Association Between HLA Gene Polymorphism and the Genetic Susceptibility of SARS Infection — https://www.researchgate.net/publication/300723620_Association_Between_HLA_Gene_Polymorphism_and_the_Genetic_Susceptibility_of_SARS_Infection